CLINICAL TRIAL: NCT03792646
Title: Effect of Protein Supplementation on Body Composition, Muscle Strength and Postural Balance in Elderly Type II Diabetes Subjects Undergoing Resistance Training
Brief Title: Protein Supplementation: Body Composition, Muscle Strength and Postural Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diabéticos
Record Dates: First submitted 2018-11-12; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2; Protein Supplementation; Body Composition; Inflammation Biomarkers; Resistance Training
Keywords: Supplementary Feeding; Protein; Muscle strenght; Exercise; Aged
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Whey Proteins; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized prospective clinical trial, double-blind, placebo-controlled intervention
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will inject 20 grams of whey protein diluted in water after the exercise training.
  Interventions: Dietary Supplement: Whey protein; Other: Exercise training
- Placebo (Placebo Comparator): The placebo group will inject 20 grams of maltodextrin diluted in water after the exercise training.
  Interventions: Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Whey protein — Exercise training + 20g whey protein
  Arms: Experimental
Other: Exercise training — Strength exercise

SUMMARY:
Nutritional interventions witch stimulate the rate of muscle protein synthesis are relevant for the development of therapeutic strategies aimed at attenuating the loss of mass and muscle strength related to aging (sarcopenia). To aim of the study is to investigate the effect of protein supplementation on body composition, muscle activity, muscle strength and plasma concentration of inflammatory biomarkers of elderly with type II diabetic, submitted to 12 weeks of resistance training. This is an interventional, controlled, randomized, double-blind study. The population of the present study will be composed of 40 men with type 2 diabetes aged between 70 and 74 years, whose body mass index (BMI) should be between 22 and 32 kg / m2. It will be composed of patients from the Diabetes Outpatient Clinic of the Endocrinology Department at the Medical School of the University of São Paulo. Elderly subjects will be randomized into two groups (n = 20) who will undergo resistance training for 12 weeks, twice a week, and receive protein or placebo supplementation. Exercises will be performed for the large muscle groups: pectoral press, paddling, leg-press, extensor chair, gastrocnemius plantar flexions and abdominal crunches. Protein supplementation will be performed immediately after strength training by ingestion of 20 g of whey protein diluted in water. Also, immediately after training the placebo group will receive 20 g of maltodextrin diluted in water. All participants will be instructed to ingest 1.0 to 1.2 g of protein / kg of body weight per day. 24-hour food recall and food frequency questionnaires will be performed throughout the study. The following evaluations (before and after 12 weeks training) will be applied: Anthropometric: body mass, height, BMI and hip waist ratio. Functional evaluation through isokinetic dynamometry of knee extensors and flexors and a maximal repetition (1RM). Evaluation of body composition through Bioimpedance balance. Evaluation of food intake will be obtained by means of a 24-hour recall and food frequency questionnaire. All the evaluations will performed after 6 months. The training sessions will have a frequency of twice a week for 12 weeks. Eight exercises will be performed for the main muscle groups. In each exercise, 3 sets will be performed between 8 and 12 repetitions. The intensity should be between 7 - 8 and will be monitored according to Subjective Effort Perception using a scale of 0 to 10.

DETAILED DESCRIPTION:
Eligibility Criteria:

Diabetes mellitus type 2 with stable dose of medication (oral antidiabetic or insulin or combination of both) for three months or more.

Glycated hemoglobin between 6 and 8.5% Renal function assessed by MDRD above 60 ml / h AST and ALT up to 2.5 times the upper limit of the No involvement of the musculoskeletal system with pain and any type of incapacitating disease or previous surgeries.

No chronic non-communicable disease not treated properly and decompensated Renal function assessed by MDRD equal to or above 60 ml / h

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 with stable dose of medication (oral antidiabetic or insulin or combination of both) for three months or more.
* Glycated hemoglobin between 6 and 8.5%
* Renal function assessed by MDRD above 60 ml / h
* AST and ALT up to 2.5 times the upper limit of the
* No involvement of the musculoskeletal system with pain and any type of incapacitating disease or previous surgeries.
* No chronic non-communicable disease not treated properly and decompensated
* Renal function assessed by MDRD equal to or above 60 ml / h

Exclusion Criteria:

• Impossibility to conduct evaluation and training efficiently

Ages: 65 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Muscular strength (hand grip) change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  Evaluation of muscular strength improvement- hand grip strength (HGS). HGS assessment was performed using a Jamar hand dynamometer, measured in kilograms (kg), which is adopted by the American Society of Hand Therapists.
Muscular strength (peak of torque) change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  Isokinetic dynamometry will be use to determine knee extension and flexion strength using the Biodex Multi-Joint System 3 (Biodex MedicalTM, Shirley, NY, USA). The isokinetic variables used was maximum peak torque corrected for body weight (%).
Muscular strength (total work) change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  Isokinetic dynamometry will be use to determine knee extension and flexion strength using the Biodex Multi-Joint System 3 (Biodex MedicalTM, Shirley, NY, USA). The isokinetic variables used was total work (J).
Postural Balance (weight transfer) change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  The postural balance assessment (posturography) was performed on the NeuroCom Balance Master® force platform system (NeuroCom International, Inc., Clackamas, Oregon, USA). The parameter measured was the mean weight transfer. The weight transfer was the time in seconds required to voluntarily shift the COG forwards, beginning in the seated position and ending with full weight-bearing on the feet.
Postural Balance (sway velocity) change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  The postural balance assessment (posturography) was performed on the NeuroCom Balance Master® force platform system (NeuroCom International, Inc., Clackamas, Oregon, USA). The parameter measured was the center of gravity (COG) sway velocity while rising. The COG sway velocity documented the degree of control over the COG above the support base during the rising phase and for 5 seconds thereafter. Sway was expressed in degrees per second.

SECONDARY OUTCOMES:
Inflammatory biomarkers - plasma concentration change from baseline (Interleukin 6) | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise).
  Peripheral blood samples (20 mL) will be collected in tubes containing EDTA anticoagulant at the initial times and 12 weeks of treatment. The total EDTA blood will be centrifuged to obtain the plasma, which will be used to evaluate the concentration of Interleukin 6 (IL-6). IL-6 is an interleukin that acts as a proinflammatory cytokine and an anti-inflammatory miocin. The IL-6 will be measure in microliter (μl)/pictogram (pg). From the whole blood with EDTA will be performed the complete blood count.
Portable Bioelectrical Impedance change from baseline | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise) and after 6 months.
  Measure body composition, such as % body fat and fat-free mass (FFM). The total body mass and body composition will be measured using a multipolar bio-impedance scale of the brand INBODY® model 230.
Inflammatory biomarkers - plasma concentration change from baseline (Tumor necrosis factor-alpha) | This measure will be perform before and after the intervention (12 weeks muscular strenght and postural balance exercise).
  Peripheral blood samples (20 mL) will be collected in tubes containing EDTA anticoagulant at the initial times and 12 weeks of treatment. The total EDTA blood will be centrifuged to obtain the plasma, which will be used to evaluate the concentration of tumor necrosis factor (TNF) -alpha. The TNF-alfa is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. The TNF-alfa wiil be measure in microliter (μl)/pictogram (pg). From the whole blood with EDTA will be performed the complete blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Greve, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- Julia Maria DÀndrea Greve, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soares ALS, Machado-Lima A, Brech GC, Greve JMD, Dos Santos JR, Inojossa TR, Rogero MM, Salles JEN, Santarem-Sobrinho JM, Davis CL, Alonso AC. The Influence of Whey Protein on Muscle Strength, Glycemic Control and Functional Tasks in Older Adults with Type 2 Diabetes Mellitus in a Resistance Exercise Program: Randomized and Triple Blind Clinical Trial. Int J Environ Res Public Health. 2023 May 20;20(10):5891. doi: 10.3390/ijerph20105891. PMID 37239618